CLINICAL TRIAL: NCT02351102
Title: Valacyclovir to Prevent Vertical Transmission of Cytomegalovirus After Maternal Primary Infection During Pregnancy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Keren shahar-nissan, Paediatrics C ward, Schneider Children's Medical Centre of Israel, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 655-14
Record Dates: First submitted 2015-01-18; First posted 2015-01-30 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Congenital Cytomegalovirus Infection
Keywords: Congenital CMV; Congenital Cytomegalovirus
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valacyclovir (Active Comparator): Participants will receive Valacyclovir at a dose of 8g/d starting at time of proof of primary maternal CMV infection and until amniocentesis (minimum 21 weeks gestation)
  Interventions: Drug: Valacyclovir
- Placebo (Placebo Comparator): Participants will receive placebo pills (same daily amount as the intervention group) starting at time of proof of primary maternal CMV infection and until amniocentesis (minimum 21 weeks gestation)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir
  Arms: Valacyclovir
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Valacyclovir treatment, administered during pregnancy after proven primary maternal Cytomegalovirus (CMV) infection, reduces fetal transmission rates and prevents fetal injury in cases of fetal infection.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study.

Participants: Pregnant women over 18 years of age with serologically proven, primary CMV infection during the first trimester

Intervention: After informed consent and randomization, participants in the treatment group will receive Valacyclovir at a dose of 8 g/d. Participants in the control group will receive the same amount of daily pills containing placebo. Treatment will continue until amniocentesis, which will determine if the fetus was infected.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women over 18 years of age with serologically proven, primary CMV infection during the first trimester of pregnancy or periconceptionally

Exclusion Criteria:

* Patients with preexisting liver disease, renal dysfunction, bone marrow suppression or sensitivity to Acyclovir will be excluded from the study - as will patients receiving any antiviral therapy prior to the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-11; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
CMV Polymerase Chain Reaction (PCR) in amniotic fluid | minimum 21 weeks gestation
  amniocentesis will be performed no earlier than 21 weeks gestation, and at least 7 weeks after estimated seroconversion occured. Therefore, the time frame for amniocentesis is estimated between 21 weeks gestation to 28 weeks gestation

SECONDARY OUTCOMES:
Clinical evidence of symptomatic congenital CMV infection | within 1 week after delivery
  laboratory, sonographic or clinical evidence of symptomatic CMV infection present after birth

CONTACTS AND LOCATIONS:
Overall Officials: Keren Shahar-Nissan, Dr, Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Helen Schneider Hospital for Women, Petah Tikva, Israel

REFERENCES:
- [Background] Buonsenso D, Serranti D, Gargiullo L, Ceccarelli M, Ranno O, Valentini P. Congenital cytomegalovirus infection: current strategies and future perspectives. Eur Rev Med Pharmacol Sci. 2012 Jul;16(7):919-35. PMID 22953641
- [Background] Gaytant MA, Steegers EA, Semmekrot BA, Merkus HM, Galama JM. Congenital cytomegalovirus infection: review of the epidemiology and outcome. Obstet Gynecol Surv. 2002 Apr;57(4):245-56. doi: 10.1097/00006254-200204000-00024. PMID 11961482
- [Background] Ornoy A, Diav-Citrin O. Fetal effects of primary and secondary cytomegalovirus infection in pregnancy. Reprod Toxicol. 2006 May;21(4):399-409. doi: 10.1016/j.reprotox.2005.02.002. PMID 16580941
- [Background] Bodeus M, Kabamba-Mukadi B, Zech F, Hubinont C, Bernard P, Goubau P. Human cytomegalovirus in utero transmission: follow-up of 524 maternal seroconversions. J Clin Virol. 2010 Feb;47(2):201-2. doi: 10.1016/j.jcv.2009.11.009. Epub 2009 Dec 16. No abstract available. PMID 20006542
- [Result] Jacquemard F, Yamamoto M, Costa JM, Romand S, Jaqz-Aigrain E, Dejean A, Daffos F, Ville Y. Maternal administration of valaciclovir in symptomatic intrauterine cytomegalovirus infection. BJOG. 2007 Sep;114(9):1113-21. doi: 10.1111/j.1471-0528.2007.01308.x. Epub 2007 Jul 6. PMID 17617198
- [Derived] Shahar-Nissan K, Pardo J, Peled O, Krause I, Bilavsky E, Wiznitzer A, Hadar E, Amir J. Valaciclovir to prevent vertical transmission of cytomegalovirus after maternal primary infection during pregnancy: a randomised, double-blind, placebo-controlled trial. Lancet. 2020 Sep 12;396(10253):779-785. doi: 10.1016/S0140-6736(20)31868-7. PMID 32919517